CLINICAL TRIAL: NCT04318626
Title: The Influence of [18F]PMPBB3 and [18F]THK5351 PET Distribution Patterns on Post-stroke Cognitive Impairment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 201802299A0
Record Dates: First submitted 2020-03-10; First posted 2020-03-24 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Post-stroke Cognitive Impairment; Neuroinflammation
Keywords: Post-stroke cognitive impairment; PET; MRI; neuroinflammation; tau protein
MeSH Terms: conditions — Neuroinflammatory Diseases; Frontotemporal Dementia | interventions — THK5351

STUDY DESIGN:
Intervention Model Description: A. Group A: Patients with acute stroke/TIA, n=50. B. Group B: Normal control, n=30.
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PMPBB3 (Other): 1. Name: [18F] PMPBB3，[18F]1-Fluoro-3-((2-((1E,3E)-4-(6-(methylamino)pyridin-3-yl)buta-1,3-dien-1-yl)ben
  2. Dosage form: intravenous injection
  3. Dose(s): 7mCi
  4. Dosing schedule: Visit 2
  5. Mechanism of action (if known): high affinity radiotracer for the tau protein
  6. Pharmacological category：Radio pharmaceutical
  Interventions: Drug: PMPBB3; Drug: THK5351
- THK (Other): 1. Name: [18F]THK5351，(S)-6-[(3-Fluoro-2-hydroxy)propoxy]-2-(2-Methylaminopyrid-5-yl)-quinoline
  2. Dosage form: intravenous injection
  3. Dose(s): 10mCi
  4. Dosing schedule: Visit 2
  5. Mechanism of action (if known): high affinity radiotracer for the tau protein
  6. Pharmacological category：Radio pharmaceutical
  Interventions: Drug: PMPBB3; Drug: THK5351

INTERVENTIONS:
Drug: PMPBB3 — F-18 PMPBB3 PET Imaging
Drug: THK5351 — F-18 THK5351 PET Imaging

SUMMARY:
Background and objects： Neuroinflammation is an active process detectable in the earliest stages of the neurodegeneration pathway. On the other hand, significant neuroinflammation, such as reactive astrocytosis, can also be observed after cerebral ischemic injury. [18F]THK5351 can monitor the neuroinflammatory process due to its high affinity to astrogliosis, and [18F]PMPBB3 is the novel tau protein radiotracer without significant off-target binding to MAO-B. The investigators hypothesize that the neuroinflammation after acute stroke may induce the tau protein accumulation. In the current proposal, our aims are to 1) explore the interaction between neuroinflammation and tau protein accumulation in acute stroke patients by applying both the [18F]PMPBB3 and [18F]THK5351 PET images and 2) determine their influence on the longterm stroke outcome and cognitive performance.

Method： The prospective project plans to recruit 2 groups of participants: one is patients with first-ever acute stroke (Group A, n=50), and the other is healthy people as the control group (Group B, n=30). Within 3 weeks of stroke, [18F]THK5351 and [18F]PMPBB3 PET will be done for imaging cerebral neuroinflammation and tau protein distribution. Brain MRI for obtaining structural and functional information will be done within 3 weeks and 3 months after stroke. Clinical and cognitive outcome will be evaluated at week 3 and months 3 and 12. In addition, APOE genotyping and carotid ultrasound will be performed as well. By obtaining the neuroimaging information, such as severity of white matter change and infarction, cortical and hippocampal atrophy, and SUVRs of [18F]THK5351 and [18F]PMPBB3 PET, the study will be able to investigate the complex interaction between neuroinflammation and tau protein accumulation after stroke, and also evaluate their influence on structural changes, stroke outcome and cognitive performance. Group comparisons will be performed using the Chi-square test, independent t test, Mann-Whitney U test, and multiple linear regression, where appropriate.

Anticipation： In this project, the investigators will be able to identify the distribution patterns of neuroinflammation and tau protein accumulation after actue stroke. Secondly, the investigators expect that the presence of neuroinflammation and tau protein accumulation will interfere with the functional connectivity. Finally, the investigators expect that the extent of neuroinflammation and tau protein is correlated with stroke outcome and post-stroke cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria for acute stroke/TIA patients (Group A, n=50)

   * Males or females with age >= 20 years old.
   * Having acute cerebral stroke or transient ischemic attack in recent 1 month.
   * Female subjects of childbearing potential must practice effective contraception during the - Provision of signed informed consent from the subject and the subject's legally
   * The subject has an appropriate caregiver capable of accompanying the subject, if necessary.
2. Inclusion criteria for healthy controls (Group B, n = 30)

   * Males or females with age >= 20 years old
   * Without history of cerebral stroke or transient ischemic attack
   * Without history of mild cognitive impairment or dementia
   * Ability to participate in cognitive and neuroimaging assessments
   * Female subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception after the final study
   * Provision of signed informed consent

Exclusion Criteria:

1. Exclusion criteria for acute stroke/TIA patients (Group A, n = 50)

   * Presence of dementia diagnosis before the index stroke or at the initial screening
   * History of vascular MCI (VaMCI)
   * The Chinese version of the Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) score >=104 at the initial screening 45.
   * Life expectancy less than 1 year.
   * Clinically significant abnormal laboratory values.
   * Clinically significant or unstable medical or psychiatric illness.
   * Epilepsy history.
   * Cognitive impairment resulting from trauma or brain damage.
   * Substance abuse or alcoholism in the past 3 months.
   * General MRI, and / or PET exclusion criteria.
   * Pregnant or becoming pregnant during the study (as documented by pregnancy testing at screening or at any date during the study according to the PI discretion) or current breast feeding.
   * History of allergy to 18F-labelled radionucleic agents, such as [18F]PMPBB3 or [18F]THK5351.
   * Subjects having high risks for the study according to the PI discretion.
2. Exclusion criteria for healthy controls (Group B, n = 30)

   * The Chinese version of the Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) score >=104 at the initial screening 45.
   * Life expectancy less than 1 year.
   * Clinically significant abnormal laboratory values.
   * Clinically significant or unstable medical or psychiatric illness.
   * Epilepsy history.
   * Cognitive impairment resulting from trauma or brain damage.
   * Substance abuse or alcoholism in the past 3 months.
   * General MRI, and / or PET exclusion criteria.
   * Pregnant or becoming pregnant during the study (as documented by pregnancy testing at screening or at any date during the study according to the PI discretion) or current breast feeding.
   * History of allergy to 18F-labelled radionucleic agents, such as [18F]PMPBB3 or [18F]THK5351.
   * Subjects having high risks for the study according to the PI discretion.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
CDR score of cognition deteriorating group and stable group | through study completion, an average of 1 year
  The CDR is a 5-point scale (0、0.5、1、2、3) used to characterize six domains of cognitive and functional performance applicable to Alzheimer disease and related dementias: Memory, Orientation, Judgment & Problem Solving, Community Affairs, Home & Hobbies, and Personal Care. The necessary information to make each rating is obtained through a semi-structured interview of the patient and a reliable informant or collateral source (e.g., family member).
  Global score 0 = Normal、0.5 = Very Mild Dementia、1 = Mild Dementia、2 = Moderate Dementia、3 = Severe Dementia. The cognition deteriorating group is defined as CDR score declines from 0 or 0.5 at Month 3 to >=1 at Month 12. The cognition stable group is defined as CDR score remains at 0 or 0.5 at Month 12.
PET imaging positive and negative conditions | through study completion, an average of 1 year
  PET images are visually assessed by independent raters, who are nuclear medicine doctors and blinded to all clinical and diagnostic information. The raters classify each scan as 0-1 (no significant uptake)、2 (suspicious uptake)、3-4 (significant uptake). The score >= 2 is deemed as positive condition.
Correlation between Neuroimaging factors and CDR-SB condition | through study completion, an average of 1 year
  Neuroimaging continuous variables will be first examined for their collinearity, determined as variance inflation factor (VIF) of 2 or more. The approach suggested by Zuur et al is to calculate VIFs for each parameter in the model, and if they are larger than some cutoff, sequentially drop the predictor with the largest VIF, recalculate, and repeat until all values are below the cutoff of 2^68. Variables showing moderate to significant inter-group difference (P < 0.10) will be selected for the logistic regression analysis (CDR-SB increase > 1 and conversion to dementia as the dependent variables).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Chang-Gung memorial Hospital, Taoyuan District, Guishan, Taiwan